CLINICAL TRIAL: NCT06442059
Title: Examination of the Relationship Between Clinical Variables and Dyspnea and Fear of Movement in Chronic Obstructive Pulmonary Patients
Brief Title: Clinical Variables and Dyspnea and Fear of Movement in Chronic Obstructive Pulmonary Patients
Status: Completed | Type: Observational
Sponsor: Kırıkkale University (Other)
Responsible Party: Principal Investigator, Saniye Aydoğan Arslan, assoc. prof. Dr., Kırıkkale University
Other Study IDs: Kırıkkaleu-Caglanyetim
Record Dates: First submitted 2024-05-29; First posted 2024-06-04 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2024-11

CONDITIONS: COPD; Kinesiophobia Due to Dyspnea
Keywords: Chronic obstructive pulmonary disease, kinesiophobia, physical performance, dyspnea
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Kinesiophobia; Dyspnea

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- copd: Patients over the age of 45 who have been diagnosed with COPD and whose clinical condition is stable
  Interventions: Other: Kinesiophobia Level Due to Dyspnea

INTERVENTIONS:
Other: Kinesiophobia Level Due to Dyspnea — Kinesiophobia Level Due to Dyspnea

SUMMARY:
Patients diagnosed with COPD who applied to the Pulmonary Diseases Department of Kırıkkale Yüksek İhtisas Hospital will be included in the study. The aim of our study: It is aimed to investigate the effect of fear of movement due to dyspnea on respiratory function, muscle strength, physical performance and balance in Chronic Obstructive Pulmonary Disease Patients.

DETAILED DESCRIPTION:
At Kırıkkale Yüksek İhtisas Hospital, individuals with COPD who meet the inclusion and exclusion criteria and volunteer to participate in the study will be included. The number of patients to be included in our study will be determined by power analysis.

Sociodemographic information (Age, Gender, Body Mass Index, Smoking history) of the individuals included in the research will be recorded.

Regarding COPD symptoms:

Whether the cough is productive or non-productive, its frequency and period Presence of sputum, type, amount, color, presence of hemoptysis, Presence of chest pain, Presence of peripheral edema, You will be asked about the presence of resting and/or exertional dyspnea, orthopnea, paroxysmal nocturnal dyspnea (PND).

1. Respiratory Muscle Strength: It will be measured using an electronic, mobile, intraoral pressure measuring device.
2. Peripheral Muscle Strength Evaluation: Quadriceps muscle strength will be evaluated using a dynomometer.
3. Physical Performance: A 6-minute walk test will be used to determine the physical fitness levels of individuals.
4. Balance Level: Mini-BEST Test will be used to determine the balance level
5. Kinesiophobia Level Due to Dyspnea:

It will be evaluated with the Breathlessness Beliefs Questionnaire (BBQ). When the literature was examined, no study was found that examined all of these factors together in patients with COPD. Existing studies have shown that the effects of variables are different and it is stated that more studies are needed.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with COPD Be clinically stable for the last four weeks Not using antibiotics for the last four weeks being over 45 years old, Volunteering to participate in the study

Exclusion Criteria:

* Not being able to cooperate with the evaluations to be made, Having any physical disability that may affect walking and balance Having severe neuromuscular, musculoskeletal and rheumatological problems accompanying COPD

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: At Kırıkkale Yüksek İhtisas Hospital, individuals with COPD who meet the inclusion and exclusion criteria and volunteer to participate in the study will be included.
Sampling Method: Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Kinesiophobia Level Due to Dyspnea | 12 moon
  It will be evaluated with the Breathlessness Beliefs Questionnaire (BBQ).BBQ; It is a scale consisting of 11 questions that evaluates the person's kinesiophobia and anxiety due to breathlessness. Patients give scores to each question ranging from 1 (strongly disagree) to 5 (strongly agree). High scores indicate high levels of kinesiophobia and anxiety due to breathlessness.

CONTACTS AND LOCATIONS:
Locations (1):
- Saniye Aydoğan Arslan, Kırıkkale, Kırıkkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided